CLINICAL TRIAL: NCT04520919
Title: Feasibility Study of a Hemodynamic Parameter Algorithm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-001
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anesthesia;Radial artery puncture — we chose the patients who need to monitor invasive blood pressure to obtain high-fidelity arterial waveforms

SUMMARY:
An algorithm to calculate hemodynamic parameters based on blood pressure waveform was developed by collecting arterial blood pressure of patients during surgery

ELIGIBILITY:
Inclusion Criteria:

* surgery patients

Exclusion Criteria:

* Weight ≤18kg arrhythmology cardiac disfunction

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who need surgery
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
arterial blood pressure | 30min~1 hour
  a high-fidelity blood pressure waveforms

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China